CLINICAL TRIAL: NCT06649812
Title: A Phase 2 Study of Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, and Revlimid (ViPOR) in Relapsed or Refractory CD10-Negative Diffuse-Large B-Cell Lymphoma (DLBCL) and High-Grade B-Cell Lymphoma With MYC and BCL2 Rearrangements (HGBCL-DH-BCL2)
Brief Title: Testing the Effectiveness of a Combination Targeted Therapy (ViPOR) for Patients With Relapsed and/or Refractory Aggressive B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-08642; NCI-2024-08642 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA4231 (Other: ECOG-ACRIN Cancer Research Group); EA4231 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: High Grade B-Cell Lymphoma With MYC and BCL6 Rearrangements; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma Germinal Center B-Cell Type; Recurrent Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Recurrent High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Recurrent High Grade B-Cell Lymphoma, Not Otherwise Specified; Recurrent T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma Germinal Center B-Cell Type; Refractory Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Refractory High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Refractory High Grade B-Cell Lymphoma, Not Otherwise Specified; Refractory T-Cell/Histiocyte-Rich Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Biopsy; Specimen Handling; ibrutinib; Lenalidomide; Magnetic Resonance Spectroscopy; obinutuzumab; Prednisone; deltacortene; prednylidene; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ViPOR) (Experimental): Patients receive venetoclax PO QD on days 2-14, ibrutinib PO QD on days 1-14, prednisone PO QD on days 1-7, obinutuzumab IV on days 1 and 2, and Revlimid PO QD on days 1-14 of each cycle. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, PET, CT and/or MRI and optional tumor biopsy and bone marrow aspiration and biopsy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Ibrutinib; Drug: Lenalidomide; Procedure: Magnetic Resonance Imaging; Biological: Obinutuzumab; Procedure: Positron Emission Tomography; Drug: Prednisone; Drug: Venetoclax

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo optional tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA 101; GA-101; GA101; Gazyva; huMAB(CD20); R 7159; R-7159; R7159; RO 5072759; RO-5072759; RO5072759
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial tests how well venetoclax, ibrutinib, prednisone, obinutuzumab, and Revlimid® (ViPOR) works in treating patients with CD10 negative diffuse large B-cell lymphoma (DLBCL) and high-grade lymphoma with MYC and BCL2 rearrangements that has come back after a period of improvement (relapsed) and/or that has not responded to previous treatment (refractory). Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Ibrutinib is in a class of medications called kinase inhibitors. It blocks a protein called BTK, which is present on B-cell (a type of white blood cells) cancers at abnormal levels. This may help keep cancer cells from growing and spreading. Anti-inflammatory drugs, such as prednisone lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Obinutuzumab, a monoclonal antibody, binds to a protein called CD20, which is found on B cells and some types of leukemia and lymphoma cells. Obinutuzumab may block CD20 and help the immune system kill cancer cells. Revlimid, a type of anti-angiogenesis agent and a type of immunomodulating agent, may help the immune system kill abnormal blood cells or cancer cells. It may also prevent the growth of new blood vessels that cancers need to grow. ViPOR may be an effective treatment option for patients with relapsed and/or refractory CD10 negative DLBCL and high-grade B-cell lymphoma with MYC and BCL2 rearrangements.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the complete response (CR) rate of ViPOR in relapsed/refractory (R/R):

Ia. CD10-negative DLBCL; and Ib. CD10-positive or negative high-grade B-cell lymphoma (HGBCL) with MYC and BCL2 (with or without BCL6) translocations (HGBCL-double hit [DH]-BCL2).

SECONDARY OBJECTIVES:

I. To evaluate the complete response (CR) rate of ViPOR in relapsed/refractory (R/R):

Ia. CD10-negative activated B-cell (ABC) DLBCL; and Ib. CD10-negative non-ABC (i.e., unclassified or germinal center B-cell [GCB]) DLBCL.

II. To evaluate the overall response rate (ORR), duration of response (DOR), event-free survival (EFS), time to progression (TTP), progression-free survival (PFS), overall survival (OS), and the safety & toxicity profile of ViPOR in relapsed/refractory (R/R):

IIa. CD10-negative ABC DLBCL; and IIb. CD10-negative non-ABC (i.e., unclassified or GCB) DLBCL; and IIc. CD10-positive or negative HGBCL-DH-BCL2.

EXPLORATORY OBJECTIVES:

I. To assess response and outcome to ViPOR based on molecular DLBCL subtype by cell-of-origin (COO) testing using Lymph2Cx gene-expression profiling (GEP).

II. To assess response and outcome to ViPOR based on genetic DLBCL subtype by LymphGen classification using whole exome sequencing (WES), whole genome sequencing (WGS), and ribonucleic acid (RNA)-sequencing (RNA-seq).

III. To determine other molecular correlates of response or resistance to ViPOR therapy.

IV. To determine early molecular correlates of response or resistance as well as the rate of complete molecular remission, as determined by assays for circulating-tumor deoxyribonucleic acid (DNA) (ctDNA).

OUTLINE:

Patients receive venetoclax orally (PO) once daily (QD) on days 2-14, ibrutinib PO QD on days 1-14, prednisone PO QD on days 1-7, obinutuzumab intravenously (IV) on days 1 and 2, and lenalidomide (Revlimid) PO QD on days 1-14 of each cycle. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, positron emission tomography (PET), computed tomography (CT) and/or magnetic resonance imaging (MRI) and optional tumor biopsy and bone marrow aspiration and biopsy throughout the study.

After completion of study treatment, patients are followed up every 6 months for 2 years, yearly during years 3-5, and then for survival for up to 10 years from the date of registration.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 18 years of age
* Patient must have histologically or cytologically confirmed aggressive B-cell lymphoma as follows:

  * Cohort 1: CD10-negative DLBCL, which includes:

    * CD10-negative non-GCB DLBCL, not otherwise specified (NOS) (i.e., CD10-/BCL6- or CD10-/BCL6+/MUM1+ DLBCL)
    * CD10-negative GCB DLBCL, NOS (i.e., CD10-/BCL6+/MUM1- DLBCL)
    * CD10-negative HGBCL with MYC and BCL6 (without BCL2) translocations (HGBCL-DH-BCL6)
    * CD10-negative HGBCL, NOS (without MYC and BCL2 translocations)
    * CD10-negative T-cell/histiocyte-rich large B-cell lymphoma (THRLBCL) OR
  * Cohort 2: CD10-positive or negative HGBCL with MYC and BCL2 rearrangements (with or without BCL6 rearrangement) (HGBCL-DH-BCL2)

    * NOTE: The site principal investigator must review and verify the pathology report findings to ensure the patient is eligible and is assigned to the respective cohort at the time of registration
* Patient must have relapsed and/or refractory disease after at least 1 prior anthracycline and anti-CD20 antibody-containing regimen
* Patient must not have confirmed or suspected primary mediastinal large B-cell lymphoma (PMBL)
* Patient must not be pregnant due to the potential harm to an unborn fetus with the treatment regimens being used.

  * All patients of childbearing potential must have a serum or urine study with a sensitivity of at least 25 mIU/mL within 14 days prior to registration to rule out pregnancy and again within 24 hours prior to starting cycle 1 day 1 of treatment.
  * A patient of childbearing potential is defined as anyone, regardless of whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patients of childbearing potential must not expect to conceive children by abstaining from sexual intercourse or by using accepted and effective methods of contraception throughout the entire duration of protocol treatment, including during dose interruptions, and for 6 months after the last dose of protocol treatment. Male patients must not father children by abstaining from sexual intercourse or by using a condom during sexual contact with pregnant partners or partners of childbearing potential throughout the entire duration of protocol treatment, including dose interruptions, and for 6 months after the last dose of protocol treatment even if they have had a successful vasectomy
* Male patients must agree to not donate semen or sperm during the entire duration of protocol treatment or for at least 28 days after the last dose of lenalidomide
* Patient must agree to abstain from breastfeeding during the entire duration of protocol treatment and for at least 6 months after the last dose of protocol treatment
* Patient must agree to abstain from donating blood during the entire duration of protocol treatment and for at least 28 days after the last dose of lenalidomide
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Absolute neutrophil count (ANC) ≥ 1,000/mcL without requirement for granulocyte colony stimulating factor (G-CSF) support (obtained ≤ 7 days prior to registration)
* Hemoglobin ≥ 8 g/dL (obtained ≤ 7 days prior to registration)
* Platelets ≥ 75,000/mcL without requirement for platelet transfusion support (obtained ≤ 7 days prior to registration)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (or ≤ 3.0 x institutional ULN for patients with documented Gilberts syndrome) (obtained ≤ 7 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3.0 x institutional ULN (obtained ≤ 7 days prior to registration)
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 30 mL/min/1.73 m^2 (estimated by Cockcroft-Gault method or measured) (obtained ≤ 7 days prior to registration)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patient must not have confirmed or suspected primary DLBCL of the central nervous system (CNS) (PCNSL)
* Patients with history of secondary CNS lymphoma (SCNSL) are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patient must not have taken or require warfarin or other strong CYP3A inhibitors or inducers within 7 days prior to registration.

  * NOTE: Antiplatelet agents, other anticoagulants aside from warfarin, as well as mild or moderate CYP3A inhibitors or inducers are permitted on study but should be used with caution
* Patient must not have an uncontrolled intercurrent illness that would interfere with the safety or efficacy assessment of this protocol
* Patient must not have evidence of an active infection at the time of registration
* Patient must not have the following current or prior anti-cancer treatment:

  * Any chemotherapy, targeted therapy, anti-cancer antibodies, antibody-drug conjugates, or bi-specific antibodies received within 2 weeks prior to registration

    * NOTE: Short courses of corticosteroids or palliative external beam radiation therapy (XRT) prior to registration are permitted
  * More than 3 prior lines of cytotoxic chemotherapy, excluding targeted therapy, anti-cancer antibodies, antibody-drug conjugates, bi-specific antibodies, and radio- or toxin-immunoconjugates

    * NOTE: Cytoreductive chemotherapy followed by autologous stem cell transplant (ASCT) counts as 1 line of cytotoxic therapy. Similarly, cytoreductive chemotherapy (either pre-T-cell collection or as bridging therapy) followed by pre-conditioning therapy/chimeric antigen receptor T-cell (CAR-T) counts as 1 line of therapy, as long as no disease progression occurs between interventions. For both therapies, if progressive disease is documented between 2 distinct regimens, then they should be counted as 2 lines of cytotoxic chemotherapy
  * Radio- or toxin-immunoconjugates within 10 weeks prior to registration
  * Previous treatment with more than one of the following study agents: venetoclax, ibrutinib, or lenalidomide
  * Prior autologous stem cell transplant (ASCT), chimeric antigen receptor T-cell (CAR-T) therapy, or allogeneic stem cell (or other organ) transplant within 3 months prior to registration
  * Any evidence of active graft-versus-host disease or requirement for immunosuppressants within 28 days prior to registration

    * NOTE: In addition, patient must have recovered (i.e., ≤ grade 1 or baseline) from all adverse events due to previously administered anti-cancer treatment, surgery, or procedure
    * NOTE: Exceptions to this include events not considered to place the patient at unacceptable risk of participation in the opinion of the treating investigator (i.e., alopecia)
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patient must have adequate formalin fixed paraffin embedded (FFPE) tumor tissue specimen from the initial diagnostic biopsy or on-study repeat tumor tissue biopsy for molecular analysis

  * NOTE: Excisional tumor biopsy is preferred. Core needle biopsies will be considered adequate if there is enough tissue for the mandatory molecular analysis. Submission of an entire FFPE tumor block is preferred, but if unavailable 10 x 10um FFPE scrolls may be submitted as an alternative. If adequate archived FFPE tumor tissue is unavailable, the patient must be willing to undergo research biopsy for molecular analysis
* Patient must have measurable disease
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate (CD10-negative diffuse large B cell lymphoma [DLBCL] and high grade B-cell lymphoma with MYC and BCL2 with or without BCL6 rearrangements [HGBCL-DH-BCL2]) | Up to 5 years
  Will be assessed using the Lugano Classification and will be defined as the complete disappearance of all detectable clinical evidence of disease, and disease-related symptoms if present prior to therapy.

SECONDARY OUTCOMES:
CR rate (CD10-negative activated B-cell [ABC] and non-ABC DLBCL) | Up to 5 years
  Estimates will be presented with 90% confidence intervals. Frequency and proportion will be used to describe variables on the nominal/ordinal scale, and measures of dispersion for interval/ratio variables. Logistic/linear regression will be performed for binary/continuous endpoints variables.
Overall response rate | Up to 5 years
  Estimates will be presented with 90% confidence intervals. Frequency and proportion will be used to describe variables on the nominal/ordinal scale, and measures of dispersion for interval/ratio variables. Logistic/linear regression will be performed for binary/continuous endpoints variables.
Duration of response (DOR) | From the documented beginning of response to the time of relapse up to 10 years
  Estimates will be presented with 90% confidence intervals. Kaplan-Meier method will be used to visualize DOR. Frequency and proportion will be used to describe variables on the nominal/ordinal scale, and measures of dispersion for interval/ratio variables. Logistic/linear regression will be performed for binary/continuous endpoints variables.
Event-free survival (EFS) | From study entry to any treatment failure including discontinuation of treatment for any reason, such as disease progression, toxicity, patient preference, initiation of new treatment without documented progression, or death up to 10 years
  Estimates will be presented with 90% confidence intervals. Kaplan-Meier method will be used to visualize EFS. Frequency and proportion will be used to describe variables on the nominal/ordinal scale, and measures of dispersion for interval/ratio variables. Multivariable analysis will be performed with Cox PH model and logistic/linear regression will be performed for binary/continuous endpoints variables.
Time of progression (TTP) | From study entry until lymphoma progression or death due to lymphoma up to 10 years
  Estimates will be presented with 90% confidence intervals. Kaplan-Meier method will be used to visualize TTP. Frequency and proportion will be used to describe variables on the nominal/ordinal scale, and measures of dispersion for interval/ratio variables. Multivariable analysis will be performed with Cox PH model and logistic/linear regression will be performed for binary/continuous endpoints variables.
Progression-free survival (PFS) | From entry onto study until lymphoma progression or death from any cause up to 10 years
  Estimates will be presented with 90% confidence intervals. Kaplan-Meier method will be used to visualize PFS. Frequency and proportion will be used to describe variables on the nominal/ordinal scale, and measures of dispersion for interval/ratio variables. Logistic/linear regression will be performed for binary/continuous endpoints variables.
Overall survival (OS) | From date of study entry to date of death up to 10 years
  Estimates will be presented with 90% confidence intervals. Kaplan-Meier method will be used to visualize OS. Frequency and proportion will be used to describe variables on the nominal/ordinal scale, and measures of dispersion for interval/ratio variables. Logistic/linear regression will be performed for binary/continuous endpoints variables.
Incidence of adverse events for patients who are CD10-negative ABC DLBCL, and CD10-negative non-ABC (i.e., unclassified or germinal center B-cell) DLBCL, and CD10-positive or negative HGBCL-DH-BCL2 | Up to 30 days after last dose of study treatment
  Toxicity data will be pooled for tabulation and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Melani, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (66):
- United States (66):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Yale University, New Haven, Connecticut
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Froedtert and MCW Moorland Reserve Health Center, New Berlin, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm